CLINICAL TRIAL: NCT05608512
Title: Emotional Labour, Mental Labour, Self-efficacy and Potential Influencing Factors of Hospice Care Nurses During COVID-19: A Mixed-method Study
Brief Title: Emotional Labor, Physical Labor and Mental Labor of Hospice Care Nurses: A Mixed-method Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Huichao Zhang, Professor, Nanjing University of Traditional Chinese Medicine
Other Study IDs: NMU22_1101
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Hospitalism
Keywords: hospice; advanced cancer; palliative care; nurse
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hospice care nurses: nurses who have worked in a palliative care or hospice unit
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — The first phase included a qualitative study. We conducted a qualitative phenomenological method to better explicate and understand palliative care nurses' emotional labor experiences, as well as the dilemmas and solutions they encounter when physical, mental, and emotional labor intertwine at work. In the early stage, we compiled an interview outline by a written qualitative meta-analysis about the emotional labor, and added the contents in the interview outline according to the actual situation in the later interview process.

SUMMARY:
Hospice care is a nurse-led multidisciplinary team care that provides physical, mental, and social care to end-of-life patients. According to the WHO, the role of hospice nurses is addressing suffering involves taking care of issues beyond physical symptoms, to support patients and their caregivers. Different from other disease care, hospice nurses face end-of-life patients and their families. As the primary nursing contact of a dying family, hospice nurses have a more intense and complex emotional experience. In China, with the improvement of human rights protection awareness, the nurse-patient relationship is particularly important, and the social requirements for nursing workers are also getting higher and higher. In addition, hospice nurses not only provide physical and psychological care to patients, but also provide comprehensive care to families of end-of-life patients. It is not just the mental work of learning expertise and dealing with emergency situations, and the physical labor of caring for large numbers of patients; but also requires emotional labor that has rarely been recognized before. When facing end-of-life patients and their families, it is particularly important to express appropriate emotions and pay emotional labor.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were nurses working as registered nurses for 6 months or more.

Exclusion Criteria:

* Nurses who were not directly involved in patient care (e.g., central sterile supply department nurses), and intern nurses were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nurses working as registered nurses for 6 months or more.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Chinese version scale of emotional labor | 1 day
  The ELS for nurses was developed by Hong and Kim (Hong & Kim, 2018), which is a 16-item scale using a five-point Likert scale ranging from 1 (not at all) to 5 (very true), with a total score ranging from 16 to 80. Higher scores indicate higher levels of emotional labor.
Depression, Anxiety, and Stress Scale -21 (DASS-21) | 1 day
  Chinese version of DASS-21 has a total of 21 items and measures three negative emotional experiences of depression, anxiety and stress (Jiang et al., 2021).

CONTACTS AND LOCATIONS:
Locations (1):
- Wu Ye, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No